CLINICAL TRIAL: NCT00914121
Title: A Single Dose, Crossover, Placebo- and Moxifloxacin- Controlled Study of the Effects of Bosutinib on Cardiac Repolarization in Healthy Adult Subjects
Brief Title: Study Evaluating The Effect of Bosutinib (SKI-606) On Cardiac Repolarization (Rhythms Of The Heart)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 3160A4-105
Record Dates: First submitted 2009-05-28; First posted 2009-06-04 (Estimated); Last update posted 2009-09-02 (Estimated); Status verified 2009-09

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — bosutinib; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- 1 (Experimental): SKI-606 alone
  Interventions: Drug: SKI-606
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- 3 (Active Comparator): Moxifloxacin
  Interventions: Drug: Moxifloxacin
- 4 (Experimental): SKI-606 plus ketoconazole
  Interventions: Drug: SKI-606
- 5 (Placebo Comparator): Placebo plus ketoconazole
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SKI-606
  Other Names: Bosutinib
  Arms: 1; 4
Drug: Placebo
  Arms: 2; 5
Drug: Moxifloxacin
  Arms: 3

SUMMARY:
The purpose of this study is to examine the effect of SKI-606 on rhythms of the heart (cardiac repolarization)

ELIGIBILITY:
Inclusion Criteria: Men or women of nonchildbearing potential; 18-50 years old; healthy as determined by the investigator, including physical examination, laboratory test results, and medical history.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-06; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Corrected QT interval, including QTcN, QTcB, and QTcF | 6 weeks

SECONDARY OUTCOMES:
Laboratory evaluations, Vital Sign measurements, Adverse Event reports | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- Tacoma, Washington, United States